CLINICAL TRIAL: NCT02251795
Title: Effects of Steady State Tipranavir/Ritonavir or Darunavir/Ritonavir or Ritonavir on Platelet Function, Coagulation and Fibrinolysis Biomarkers in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.117
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Darunavir; Aspirin

ARMS (3):
- Tipranavir/Ritonavir (Experimental): 500 mg Tipranavir / 200 mg Ritonavir 10 days BID
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Aspirin
- Darunavir/Ritonavir (Active Comparator): 600 mg Darunavir /100 mg Ritonavir 10 days BID
  Interventions: Drug: Ritonavir; Drug: Darunavir; Drug: Aspirin
- Ritonavir (Active Comparator): 100 mg Ritonavir 10 days BID
  Interventions: Drug: Ritonavir; Drug: Aspirin

INTERVENTIONS:
Drug: Tipranavir
  Other Names: APTIVUS®
  Arms: Tipranavir/Ritonavir
Drug: Ritonavir
  Other Names: Norvir®
Drug: Darunavir
  Other Names: PREZISTA®
  Arms: Darunavir/Ritonavir
Drug: Aspirin — single dose on day 2
  Other Names: Acetylsalicylic acid

SUMMARY:
Study to determine the effect of steady-state plasma concentration of Tipranavir/ritonavir (TPV/r) on platelet aggregation in healthy subjects and investigate the effect of TPV/r at steady state plasma concentrations on other platelet functions and biomarkers of coagulation and fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give written informed consent to participate in this study (i.e., prior to any study-specific procedures)
2. Age ≥18 years and ≤50 years
3. Female subjects of child-bearing potential were eligible if:

   * They had used a barrier contraceptive method for at least 12 weeks before administration of study medication and had a negative serum pregnancy test result during the screening period (Day - 35 to Day -3); or,
   * Were abstinent for more than 12 weeks before screening and had a negative serum pregnancy test result during the screening period (Day -35 to Day -3); or,
   * Had a documented tubal ligation and had a negative serum pregnancy test result during the screening period (Day -35 to Day -3)
4. Ability to swallow capsules without difficulty
5. Reasonable probability of completing the study
6. Findings from medical history, physical examination and 12-lead ECG indicating subject was healthy and suitable for the trial in the opinion of the investigator
7. Agreement to abstain from alcohol consumption or drugs of abuse during the study
8. Agreement to abstain from ingestion of grapefruit, grapefruit juice, Seville oranges, or orange marmalade from screening period to the end of the study
9. Negative urine drug screen for drugs of abuse
10. Non smoker
11. Agreement to abstain from use of tobacco products from screening period to the end of the study
12. Negative HIV-1 serology by ELISA testing
13. Negative Hepatitis B surface Antigen test (HBsAg)
14. Negative Hepatitis C Virus antibody (anti-HCV) test by Enzyme Immunoassay
15. Platelet count ≥125,000/mm3
16. Hemoglobin ≥11.0 g/dL
17. Prothrombin time ≤1.0 x upper limit of normal (ULN)
18. Activated Partial thromboplastin time ≤1.0 x ULN

Exclusion Criteria:

1. Female subjects who:

   * had a positive serum pregnancy test during the screening period (Day -35 to Day -3) or during the study
   * were breast feeding or planing to breast feed at any time from the screening period through 30 days after the last dose of the study drug
   * were not willing to use a barrier method of contraception at any time from screening period through 30 days after the last dose of the study drug
   * were taking any hormonal therapy for any reason such as birth control or replacement therapy
2. Had used any investigational agent within 30 days prior to Visit 2
3. Blood or plasma donations (>100 mL total) for research or altruistic reasons within 30 days prior to Visit 2
4. Had used aspirin or any non-steroidal anti-inflammatory agent (NSAID), and including COX-2 inhibitors, dipyridamole, clopidogrel, ticlopidine or other antiplatelet drugs within 14 days prior to Visit 2 or during the study
5. Active peptic ulceration or history of peptic ulcer disease
6. Known history of or suspected hypersensitivity to aspirin, any NSAID or any other component of the test drugs (Tipranavir, Darunavir, Ritonavir)
7. Known hypersensitivity to antiretroviral drugs (marketed or experimental drug in clinical research studies)
8. Active bleeding disorder or history of active bleeding disorder
9. Active Intra cranial hemorrhage (ICH) or history of ICH
10. Active coronary artery disease or history of coronary artery disease
11. Alcohol abuse (more than 60 g/day)
12. Any indication for current use of aspirin or any NSAID or indication for such use from Visit 2 to Visit 18
13. Had used any over-the-counter medication within 7 days prior to Visit 2, or current use of any prescription drug
14. Subjects who had an abnormal laboratory result of Grade 1 or greater, as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS), (result must have been available at least 3 days prior to Visit 2-Day 1), except the following screening laboratory values:

    * serum potassium, serum sodium, serum phosphate and uric acid, where central laboratory reference ranges will be used to determine eligibility rather than DAIDS table; or,
    * amylase or creatinine results of Grade 1 on DAIDS table if these results are considered clinically not significant by investigator; or
    * other marginally abnormal laboratory values not considered clinically significant by investigator and approved by clinical monitor
15. History of any illness that in the opinion of the investigator might confound the results of the study or pose additional risks in administering aspirin, Tipranavir, Darunavir, or Ritonavir
16. Hypersensitivity to sulphonamide drugs
17. Had used proton pump inhibitors during 14 days prior to Visit 2
18. Vitamin E intake in excess of 60 mg/day within 30 days prior to Visit 2
19. Vitamin E supplementation in excess of 60 mg/day during the study (Vitamin E content of multivitamin tablets is allowed)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in the area under the curve (AUC) of platelet aggregation in response to arachidonic acid (AA) | pre-dose, up to 48 h after drug administration
  calculated as the ratio of the AUC at steady state TPV plasma concentrations and the baseline AUC

SECONDARY OUTCOMES:
Changes in platelet aggregation in response to AA | pre-dose, up to 48 h after drug administration
Changes in platelet aggregation in response to collagen | pre-dose, up to 48 h after drug administration
Changes in platelet aggregation in response adenosine diphosphate (ADP) | pre-dose, up to 48 h after drug administration
Changes in closure Time (CT) | pre-dose, up to 48 h after drug administration
  Platelet Function Analyzer (PFA)-100 test
Changes in urinary thromboxane B2 metabolites | pre-dose, up to 48 h after drug administration
Changes in bleeding time | Baseline, up to day 30
Changes in activated partial thromboplastin time (aPTT) | Baseline, up to day 30
Changes in prothrombin time (PT) | Baseline, up to day 30
Changes in fibrinogen | Baseline, up to day 30
Changes in von Willebrand antigen | Baseline, up to day 30
Changes in von anti-thrombin III antigen | Baseline, up to day 30
Changes in anti-thrombin III activity | Baseline, up to day 30
Changes in factor II | Baseline, up to day 30
Changes in factor VII | Baseline, up to day 30
Changes in factor IX | Baseline, up to day 30
Changes in factor X | Baseline, up to day 30
Changes in plasminogen activity | Baseline, up to day 30
Changes in alpha 2-antiplasmin | Baseline, up to day 30
Changes in D-dimer | Baseline, up to day 30
Changes in Plasminogen Activator Inhibitor (PAI-1) | Baseline, up to day 30
Maximum measured concentration of the analyte in plasma (Cmax) | pre-dose, up to 48 h after drug administration
Serum concentration at 12 hours (Cp12h) | 12 hours after drug administration
Area under the curve from 0-12 hours (AUC0-12h) | up to 12 hours after drug administration
Time from dosing to the maximum measured concentration of the analyte in plasma (Tmax) | up to 48 h after drug administration
Total clearance of the analyte in plasma (CL/F) | pre-dose, up to 48 h after drug administration
Apparent volume of distribution (V/F) | pre-dose, up to 48 h after drug administration
Terminal half-life (t1/2) | pre-dose, up to 48 h after drug administration
Number of subjects with abnormal findings in laboratory tests | up to day 61
Number of subjects with treatment-emergent adverse events | up to 96 days